CLINICAL TRIAL: NCT02021175
Title: Adaptation and Development of a Web and Cell Phone Quit Smoking Treatment for Korean Youth
Brief Title: Korean Youth Smoking Cessation Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to build the app for the clinical trial
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P60MD006923 (NIH); P60MD006923 (NIH)
Record Dates: First submitted 2013-02-06; First posted 2013-12-27 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Smoking Cessation; Korean; Youth; Adolescent; Dependence; Teen Smoking; Smoking and Youth; Youth and Tobacco; Cognitive-Behavioral Motivational Enhancement; Technology; Nicotine Dependence; Cell Phone; Smart Phone; Internet; Web
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored CBME Therapy via Technology (Experimental): 6 weeks of tailored interactive Cognitive-Behavioral Motivational Enhancement Therapy delivered through internet and cell phones
  Interventions: Behavioral: Tailored CBME Therapy via Technology
- Standard of Care (Other): Referral to currently available resources for 6 weeks of a standard smoking cessation approach
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Tailored CBME Therapy via Technology — 6 Sessions of tailored interactive Cognitive-Behavioral Motivational Enhancement Therapy delivered through internet and cell phones
  Arms: Tailored CBME Therapy via Technology
Other: Standard of Care — Referral to currently available resources for 6 sessions of a standard smoking cessation approach
  Arms: Standard of Care

SUMMARY:
Cigarette smoking remains the leading preventable cause of morbidity and mortality in the United States. In Los Angeles, rates of morbidities due to cigarette smoking follow prevalence. While the rate of cigarette smoking in Los Angeles County among youth is at historic lows, prevalence is not uniform: Cigarette smoking is pervasive among residents who have significant economic disparities. Prevalence is also among the highest in the world for Korean school-aged youth and substantially higher numbers of Korean American youth smoke cigarettes. To date, smoking prevention efforts in Korea have had mixed results as they are not interesting to youth and are not interactive.

This project will assess an interactive, culturally adapted, tailored smoking cessation intervention delivered through the internet and cell phone. Using technology, the investigators seek to increase the reach and access of our intervention and facilitate cessation without in-person sessions, a factor that limits smoking cessation interventions for youth. Youth are energetic users of electronic media, lending support to the delivery of treatment through technology.

The investigators predict that subjects assigned to the intervention will demonstrate statistically higher rates of smoking abstinence and longer retention in the cessation program compared to those assigned to the standard of care condition. Subjects reporting higher levels of smoking exposure, lower motivation, poor mental health, disadvantaged neighborhoods, and lower levels of acculturation to American culture will also have lower quit rates at each follow-up visit.

DETAILED DESCRIPTION:
Cigarette smoking remains the leading preventable cause of morbidity and mortality in the United States. While 19% of U.S. twelfth graders smoked cigarettes in the past 30 days, fewer than 10% of Californians under age 18 reported recent smoking. In Los Angeles, rates of morbidities due to cigarette smoking follow prevalence. While the rate of cigarette smoking in Los Angeles County among youth is at historic lows (10.4%), prevalence is not uniform: Cigarette smoking is pervasive among residents who have significant economic disparities. Alarming racial and ethnic disparities are noted with highest prevalence reported for adult Korean males (44.8%). Prevalence of cigarette smoking is also among the highest in the world for Korean school-aged youth, with 16.2% for males and 5.3% for females. To date, smoking prevention efforts in Korea have had mixed results as they are not interesting to youth and are not interactive.

This project will assess an interactive, culturally adapted, tailored smoking cessation intervention delivered through the internet and cell phone. The evidence-based treatment, "Cognitive-Behavioral/Motivational Enhancement Therapy for Smoking Cessation" (CBME) for adolescent smokers was developed by one of the investigators. Based on input from our community partners, consultants, and youth focus group participants, the treatment will be culturally adapted for appropriateness and relevance to Korean youth. The refined intervention will be programmed for delivery via the Web and mobile technologies. Using technology, we seek to increase the reach and access of our intervention and facilitate cessation without in-person sessions, a factor that limits smoking cessation interventions for youth. A 2-group, randomized control trial design will assign youth either to the tailored Web and cell phone based smoking cessation program or to a control condition.

The specific aim of the study is as follows:

1. To evaluate the efficacy of the tailored smoking cessation approach for Korean youth seeking smoking cessation, randomly assigning 240 youth to either the experimental condition or to a standard cessation approach.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Korean or Korean-American
* Smoke at least 5 cigarettes per day for the past 6 months
* Interested in smoking cessation
* Aged between 14-19 years
* Willing to provide information that can assist in locating the individual for follow up visits
* Living in Los Angeles County
* Has a phone capable of receiving Short Message Service (SMS) text messages
* Has a computer or other regular access to engage program components
* Willing and able to provide consent if older than 18
* Willing and able to provide assent if under 18 and has a parent or legal guardian willing and able to provide consent
* At least 6th grade English reading level due to requirements of assessment procedures

Exclusion Criteria:

* Knowingly moving from the Los Angeles County area in the next year
* Absence of cotinine in urine during the baseline screen
* Concurrent dependence on substance other than nicotine
* History of suicidality in the past year
* Any other circumstances that, in the opinion of the investigators, would compromise participant safety

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in 7-day point prevalence of smoking abstinence at the end of treatment and at 6-month follow-up evaluations. | 18 weeks
  At each follow up visit, 7-day point prevalence of smoking abstinence verified by urinary cotinine and carbon monoxide (CO) will be assessed. Variables that mediate outcomes include measures of demographics, withdrawal symptoms, psychiatric and substance use status, impulsivity, health-related quality of life, and neighborhood status and acculturation.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Shoptaw, Ph.D, Principal Investigator — University of California Los Angeles, Center for Behavioral and Addiction Medicine; Vickie Mays, Ph.D, Principal Investigator — University of California Los Angeles, Center for Bridging Research, Innovation, Training, and Education on Minority Disparities Solutions (BRITE)
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States